CLINICAL TRIAL: NCT00329290
Title: Evaluation of Maternal and Fetal Outcomes in Pregnancies in Women With Prosthetic Heart Valves
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 068-02
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Pregnancy; Anticoagulation; Prosthetic Heart Valves
Keywords: pregnancy; anticoagulation; enoxaparin; prosthetic heart valves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The ability to diagnose and surgically repair poorly functioning heart valves has yielded a significant population of women that are of childbearing age with mechanical/ bioprosthetic heart valves. The clinical management of pregnant women with artificial heart valves during pregnancy has been difficult. Currently there have not been any controlled clinical trials to provide guidelines for a safe and effective anticoagulation. Current review of the literature has shown that oral anticoagulation with warfarin has been implicated to cause significant fetal morbidity including prematurity, decreased birth weight, birth defects (i.e.:"warfarin embryopathy"), abortions, still birth and neonatal mortality. Warfarin embryopathy refers to characteristic anomalies (nasal hypoplasia, eye defects, hypoplasia of extremities, deafness, mental and developmental retardation), that may occur when coumadin is used during first trimester and/or if used in doses >5mg per day during pregnancy. It has also been reported that intravenous and subcutaneous heparin has not been sufficiently effective in lowering maternal morbidity and mortality. Thromboembolic events, valve dysfunction leading to peripartum valve replacements, and maternal death have all been observed.

The purpose of this study is to:

* Evaluate the outcome of pregnancy in women with mechanical/bioprosthetic heart valves.
* Identify the risks posed to both mother and fetus during treatment with various methods of anticoagulation during pregnancy.

The survey will be conducted in three phases:

Physicians who respond to:

Phase 1: A questionnaire asking physicians whether they have cared for a patient with prosthetic heart valve after year 1990 will be mailed, faxed or e-mailed to all members of the Society of Maternal Fetal Medicine.

Phase 2: Responding physicians will provide information for the investigators to contact their patients and obtain a telephone/signed consent form (approved by the LBMMC IRB) to participate in the study and release their medical records to the investigators.

Phase 3: Data will be collected by the investigators/research nurse by reviewing medical records and interviewing referring physicians and the patients.

Although the information may not have immediate benefit to the subject, the data collected may help the medical community develop a more effective guideline of selection of prosthetic valves in women in the childbearing age and care of patients with prosthetic heart valves during pregnancy.

DETAILED DESCRIPTION:
Title of Project:

Evaluation of Maternal and Fetal Outcomes in Pregnancies in Women with Prosthetic Heart Valves

Specific Aims and Purpose of this Descriptive Study

* Evaluate the outcome of pregnancy in women with mechanical/bioprosthetic heart valves.
* Identify the risks posed to both mother and fetus during treatment with various methods of anticoagulation during pregnancy.

Hypothesis and Expected Outcomes

Patients with prosthetic heart valves in pregnancy constitute an extremely high risk group with adverse maternal and perinatal outcomes. The study is expected to review and possibly guide anticoagulation issues, and the risks associated with various therapeutic options, i.e. coumadin vs. unfractionated heparin vs. low molecular weight heparin. In addition, the study will provide information and possibly suggest an optimal way to manage such patients.

Background and Significance:

The ability to diagnose and surgically repair poorly functioning heart valves has yielded a significant population of women that are of childbearing age with mechanical/ bioprosthetic heart valves. The clinical management of pregnant women with artificial heart valves during pregnancy has been difficult. Currently there have not been any controlled clinical trials to provide guidelines for a safe and effective anticoagulation. Current review of the literature has shown that oral anticoagulation with warfarin has been implicated to cause significant fetal morbidity including prematurity, decreased birth weight, birth defects (i.e.: "warfarin embryopathy"), abortions, still birth and neonatal mortality. Warfarin embryopathy refers to characteristic anomalies (nasal hypoplasia, eye defects, hypoplasia of extremities, deafness, mental and developmental retardation), that may occur when coumadin is used during first trimester and/or if used in doses >5mg per day during pregnancy. It has also been reported that intravenous and subcutaneous heparin has not been sufficiently effective in lowering maternal morbidity and mortality. Thromboembolic events, valve dysfunction leading to peripartum valve replacements, and maternal death have all been observed.

Inclusion Criteria:

* Females with prosthetic heart valve/s who became pregnant after their surgical valve replacement.
* Complete medical information (medical history, surgical history, medication history, prosthetic heart valve information, anticoagulation history, obstetrical history, delivery history, fetal outcome, complications) obtained from patients' records and/or patients' physicians.

Exclusion Criteria:

* Patients in whom sufficient information cannot be obtained from either medical records or physicians.
* Patients who do not give written consent.

Research Design and Methods:

The survey will be conducted in three phases:

Physicians who respond to:

Phase 1: A questionnaire asking physicians whether they have cared for a patient with prosthetic heart valve after year 1990 will be mailed, faxed or e-mailed to all members of the Society of Maternal Fetal Medicine.

Phase 2: Responding physicians will provide information for the investigators to contact their patients (spouse/next to kin if the patient is deceased), and obtain a telephone/signed consent form (approved by the LBMMC IRB) to participate in the study and release their medical records to the investigators.

Phase 3: Data will be collected by the investigators by reviewing medical records and interviewing referring physicians and the patients.

In the event that the patient cannot authorize informed consent due to death, lost to follow-up, or other incapacitating illness, and next of kin cannot be reached, the primary doctor will be asked to provide necessary, relevant medical records without disclosure of the patient's identity.

Parameters used for assessment of patients' demographics as well as maternal and fetal outcome are included in the enclosed form (Form 2).

Telephone interviews, if needed, will be done at the patient's convenience.

Data Storage and Confidentiality:

Research data will be stored at our office. All information that is obtained in connection with this study will remain confidential. If the results of this study are published or presented at meetings, the identity of the subjects will not be disclosed.

Potential Benefits to the Subject:

Although the information may not have immediate benefit to the patient, the data collected may help the medical community develop a more effective guideline of selection of prosthetic valves in women in the childbearing age and care of patients with prosthetic heart valves during pregnancy.

Therapeutic Alternatives:

The alternative is not to participate in this study.

Clinical Significance:

This study could provide information regarding maternal and fetal risks associated with pregnancy in women with prosthetic heart valves. This information will be useful for risk assessment prior to pregnancy as well as for management of patients during pregnancy, especially in regard to most appropriate anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Females with prosthetic heart valve/s who became pregnant after their surgical valve replacement.
* Complete medical information (medical history, surgical history, medication history, prosthetic heart valve information, anticoagulation history, obstetrical history, delivery history, fetal outcome, complications) obtained from patients' records and/or patients' physicians.

Exclusion Criteria:

* Patients in whom sufficient information cannot be obtained from either medical records or physicians.
* Patients who do not give written consent.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Questionare
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2002-02; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afshan B Hameed, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States